CLINICAL TRIAL: NCT02936427
Title: The Effects and Dose Response of Dexamethasone on Intercostal Nerve Blocks With Bupivicaine in Post Thoracic Surgery Patients
Brief Title: Effects and Dose Response of Dexamethasone on Intercostal Blocks With Bupivicaine in Post Thoracic Surgery Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Mark Murphy, Surgical SHO, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PIL/Consentvs1
Record Dates: First submitted 2016-05-21; First posted 2016-10-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Control group will receive normal post operative care including intercostal wound catheters however will not receive dexamethasone
- Dexamethasone 4mg (Experimental): Participants will receive 4mg of dexamethasone into the intercostal space surrounding the intercostal nerve prior to the first incision. They will then receive routine post operative care including intercostal wound catheters.
  Interventions: Drug: Dexamethasone
- Dexamethasone 8mg (Experimental): Participants will receive 8mg of dexamethasone into the intercostal space surrounding the intercostal nerve prior to the first incision. They will then receive routine post operative care including intercostal wound catheters.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — perineural infiltration of dexamethasone
  Other Names: Dexamethasone phosphate
  Arms: Dexamethasone 4mg; Dexamethasone 8mg

SUMMARY:
Post-op analgesia is the most important part of early and safe patient recovery in thoracic surgery. This is for both humane and patient outcome reasons. Patient outcomes are greatly improved with optimal pain control and complications and length of stay are minimized. Most post-op thoracic complications are from decreased respiratory effort, failure to clear secretions and pulmonary infections from retained sputum with subsequent sequelae. Good post-operative analgesia not only prevents these complications but also considerably enhances early mobilization and thus, decreased hospital stay and efficient resource allocation. Early post-operative pain is also associated with late and chronic post thoracotomy pain syndromes which can be debilitating.

Pain following thoracic surgery is different to the standard surgical incision pain and is due to intercostal nerve damage, compression or traction injury to the nerve. This occurs with the incision, rib retraction, and is compounded by the on-going need for respiratory effort. The approach to managing this pain is multi-modal analgesia. The standard regimen stretches from preemptive analgesia and preoperative placement of thoracic epidurals to post-op opioid infusions. However, non-invasive pharmacology includes paracetamol, non steroidal anti inflammatory drugs (NSAIDs), mild and moderate opioids as well as anti-convulsants like pregabalin. However, opioid use has well-known side effects including central nervous system (CNS) and respiratory depression which unfortunately delay mobility and recovery. This has motivated opioid-sparing strategies.

The investigators study aims to assess whether the addition of perineural dexamethasone (a steroid) to the current practice of local anaesthetic wound catheters increases the efficacy and duration of analgesia provided.

DETAILED DESCRIPTION:
Recent years have seen the importance of early mobility and respiratory toilet to minimise complications and hospital stay. Newer methods of pain relief with fewer systemic effects have become even more important. Continuous wound infiltration catheters (CWI's) aim to deliver local anaesthetic agents directly into the wound (4). This technique goes back to 1994, and has been established in this hospital and is used in a non-structured manner in thoracic surgery. Recent studies have demonstrated that the addition of dexamethasone (a steroid) to local anaesthetic agents in similar nerve blocks significantly improves the analgesic affect and prolongs the duration of the analgesia. To the best of the investigators knowledge this has not been tested in a thoracic surgery cohort of patients, though it has been tested safely and effectively in the thorax in healthy volunteers and in postoperative analgesia in abdominal and musculoskeletal post op patients. The investigators aim is to assess whether the addition of perineural dexamethasone to the local anaesthetic in CWI's is superior to the local anaesthetic alone in thoracic post operative patients, and at which dose. They also want to assess the levels of pain experienced 1 month post op to evaluate the potential effect of dexamethasone on post thoracoscopy pain syndrome.

The investigators aim is to compare the use of local anaesthetic agent in combination with perineural dexamethasone with the current practice of local anaesthetic alone at relieving pain in the immediate post op pain period. The investigators also want to assess whether the 8mg dose of dexamethasone used in similar studies is the optimal dose or whether a similar effect can be observed at a smaller dose of 4mg.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Consenting
* undergoing VATS procedure

Exclusion Criteria:

* Age <18
* Refusal to consent
* Equipment failure
* Allergic reactions to local anaesthetic agent
* Incipient agents or opioid
* Patients on pre-existing long-term opioid use
* Any other concomitant or surgery within 2 weeks of the thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Amount of analgesia used in 24hrs | 0- 24hrs from surgery
  Cumulative analgesia used over 24hrs
Amount of analgesia used in 48hrs | 0-48hrs from surgery
  Cumulative analgesia used in 48 hrs
Amount of analgesia used in 1 month from date of surgery | 0hrs - 1 month from surgery
  Cumulative analgesia used over 1 month

SECONDARY OUTCOMES:
Pain reported by patient at 24hrs | recording of patients level of pain 24hrs post op
  Pain according to Visual analog score reported by the patient
Pain reported by patient at 48hrs | recording of patients level of pain 48hrs post op
  Pain according to Visual analog score reported by the patient
Pain reported by patient 1 month post op | recording of patients level of pain 1 month post op
  Pain according to Visual analog score reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Murphy, MB BcH BAO, Principal Investigator — Surgical SHO
Locations (1):
- St Vincent's University Hospital, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided